CLINICAL TRIAL: NCT07240883
Title: ENDO1000 - A UK-wide Endometriosis Research Project
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Clinical Hospital Centre Zagreb (Other); Endometriosis UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: 101157146; 101157146 (Other Grant/Funding Number: Horizon Europe Framework Programme (HORIZON) and philanthropic donations)
Record Dates: First submitted 2025-09-05; First posted 2025-11-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis
Keywords: Endometriosis; Pelvic Pain; Longitudinal; Mobile app
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood, urine, saliva, faeces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Sample and data collection — We will collect data via a bespoke mobile application which will include; pain, fatigue, sleep patterns, diet, bowel habits, exercise, painkiller use, hormone use from participants with endometriosis. In a subset of the participants, we will collect biological samples which will be self collected at home, that will include, blood, saliva, urine and faeces. At time of sample collected, we will also ask a selection of validated questionnaires to be completed.

SUMMARY:
Approximately 1.5 million people in the UK, and 200 million globally live with endometriosis, and it is estimated to affect 1 in 10 women of reproductive age. Endometriosis is a chronic pain condition where the lining of the uterus (endometrium) grows in areas outside the uterus. This can cause patients a range of symptoms including severe pain, fatigue, irregular periods, infertility and gastrointestinal symptoms.

There is a clear unmet need for early diagnosis and more effective pain management for people who suffer from endometriosis. Endometriosis is a heterogeneous disease in terms of symptoms, trajectory, and indicated therapeutic course, which highlights the need to develop personalised/targeted approaches for effective longitudinal management which are acceptable and accessible to patients and their health care team.

The goal of this study is to accelerate discovery and advance data-driven research into endometriosis diagnosis and treatment by collecting large, multimodal, longitudinal data.

To achieve this goal, the investigators plan to deliver a longitudinal cohort study. Approximately 3000 UK individuals with endometriosis will be invited over a 24-month period to self-report symptoms that include, pain, menstrual cycle, painkiller use, sleep, exercise, diet and bowel habits via a bespoke ENDO1000 mobile app. A cohort of 1000 women will be asked to complete more in-depth questionnaires asking about endometriosis history, quality of life and treatments. This cohort of women will be asked to take self-collected biological samples (blood, urine, saliva, vaginal swab and faeces). The investigators will look at, for example, inflammatory markers, examine the microbiome and may look at DNA, with permission to see if there are any markers that can help with diagnosis or treatment of endometriosis. At the same time participants will be asked to wear a smartwatch which will monitor, for example, temperature, ambient light, sleep patterns and movement. All this will help the investigators to build a picture over time of the participant's endometriosis symptoms, treatments and what may cause symptoms to flare which in turn could lead to more patient led treatments.

DETAILED DESCRIPTION:
BACKGROUND Endometriosis is characterised by the presence of endometrial-like tissue ('lesions') outside the uterus, commonly on the lining of the pelvic cavity. It is a chronic, inflammatory gynaecological condition that affects approximately 6-10% of women and those assigned female at birth. It is associated with debilitating pelvic pain, gastrointestinal and urinary symptoms, fatigue and infertility. Endometriosis can profoundly affect quality of life, limiting daily activities, social engagement, physical and sexual health, relationships, career and educational pursuits, mental well-being, and overall health. It is associated with a 45% reduction in work productivity with an annual cost for caring for women with endometriosis estimated at > £8.2 billion per year in the UK.

People with endometriosis experience an average of 8 years of delay in the UK from the onset of their symptoms before receiving a diagnosis. There are no validated non-invasive tests for endometriosis and the current gold standard for diagnosis is via a diagnostic laparoscopy. Currently, the waiting time for this procedure in the UK is variable across NHS Trusts and can be up to two years.

Treatment options typically include:

* Painkillers e.g. paracetamol, NSAIDs.
* Surgery to remove endometriosis lesions, although this is ineffective in an estimated 30 % of women and, even when its effective, symptoms return in up to 50% of women within 5 years of surgery.
* Hormone therapies, which are not curative, can have significant side effects and are contraceptive.

Some individuals explore lifestyle changes, such as dietary adjustments or exercise, but research on the effectiveness of these approaches remains limited.

RATIONALE FOR STUDY

Endometriosis is a heterogeneous disease in terms of symptoms, trajectory, and indicated therapeutic course, which highlights the need to develop personalised and targeted approaches for effective longitudinal management which are acceptable and accessible to patients and their health care team.

There is a clear unmet need for earlier diagnosis and more effective pain management for people who suffer from the condition.

The goal of this study is to accelerate discovery and advance data-driven research into endometriosis diagnosis and treatment by collecting large, multimodal, longitudinal data. This study is for the collection of data which will be retrospectively analysed. No feedback will be given to the individual participants on the results.

To achieve this goal, the investigators plan to deliver a longitudinal cohort Approximately 3000 UK individuals with endometriosis will be invited to take part in the study. participants will be asked to do the following over a 24-month period:

1. Record information about their pain, physical functioning, mental health/emotional functioning, diet/sleep, medical/surgical interventions and self-management strategies on a bespoke smartphone app specifically developed for the needs of this project
2. Wear smartwatches for up to four, six-week periods to collect raw actigraphy data (three-dimensional acceleration, wrist temperature, ambient light) from which we can objectively infer longitudinal physical activity, sleep, and circadian variability characteristics using algorithms we have developed in-house. The smartwatches will be posted to participants and include pre-paid envelopes for their return to the research team, following similar protocols we have already developed and successfully deployed at the University of Edinburgh in related longitudinal studies (e.g. the SHAW study, https://www.shaw.business-school.ed.ac.uk/).
3. Obtain serial self-collected samples of saliva, blood, faeces and urine on up to four occasions. Sample collection kits will be sent to participants by our research team by post, self-collected at home and posted by participants back to our research team for analysis in our laboratory. This approach in collecting samples remotely will allow us to collect information from a diverse population of patients with endometriosis UK-wide and builds on our experience with longitudinal data collection.

The proposed study has been informed by those with lived experience of endometriosis and by representatives from the UK patient organisation, Endometriosis UK.

ELIGIBILITY:
INCLUSION CRITERIA

1. Aged 16 or over
2. Participants who confirm that they have received a clinical diagnosis of endometriosis (based on MRI, ultrasound or laparoscopy) within the last 10 years
3. Living within the UK
4. Willing and able to consent to installing and using the mobile ENDO1000 app on their smartphone or use our web-based equivalent.

EXCLUSION CRITERIA

1. Pregnant
2. Known severe coagulation disorder
3. Known active Hepatitis B/C and/or HIV (due to Royal Mail restrictions on biospecimen postage)

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anyone living within the UK with a self-reported diagnosis of endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To generate a unique biomedical endometriosis resource with detailed clinical and lifestyle phenotyping. | 5 years
  This study aims to characterise overall endometriosis symptom severity. This is a multifaceted objective to cover the breadth of symptoms of endometriosis and there is not a single scale that captures this that could be assigned as "primary outcome measure". We aim to define a new gold standard, on the basis of the largest longitudinal multimodal endometriosis study ever conducted. We envisage the resulting clinical score will be derived by combining different symptoms as experienced by patients and combining different data modalities.
  Specifically, we will elicit responses where participants self-quantify: pain (EHP-30), fatigue (BFI), sleep problems (PSQI and PROMIS), bowel habits (NHS questionnaire), diet (FFQ), epidemiological and genetic data (WERF EPHect Patient Questionnaire).
  Additional inputs will be provided by biological samples and data from a wrist-worn wearable sensor, from which we have validated algorithms to characterise physical activity, sleep and diurnal rhythm.

SECONDARY OUTCOMES:
To use the biomedical endometriosis resource to address fundamental questions in our understanding of endometriosis. | 5 years
  (i) To investigate the potential for patient stratification/prediction of treatment response from clinical/biological data profiles.
  (ii) To investigate the relationship between symptoms of pelvic pain and the gut-brain axis (including microbiome) using multi-omics data.
  (iii) To demonstrate longitudinal endometriosis symptom trajectories using app-based patient reported outcome measures (PROMs) and wearable technology.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Horne, PhD, MB ChB, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT07240883/Prot_000.pdf